CLINICAL TRIAL: NCT00002479
Title: Phase II Trial of Tretinoin (TRA) in Patients With Mycosis Fungoides/Sezary Syndrome
Brief Title: Tretinoin in Treating Patients With Mycosis Fungoides or Sezary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NCI T91-0136; NU-T91-0136; NCI-T91-0136O
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tretinoin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of tretinoin in treating patients who have any stage mycosis fungoides or Sezary syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of tretinoin (TRA) in patients with mycosis fungoides/Sezary syndrome. II. Evaluate the spectrum of toxicity of TRA in this patient population.

OUTLINE: Nonrandomized study. Single-agent Chemotherapy. Tretinoin, All-trans-Retinoic Acid, TRA, NSC-122758.

PROJECTED ACCRUAL: If 1 or more of the first 15 evaluable patients experience an objective response, then 20 additional patients will be entered. It is anticipated that the accrual rate will be 1-2 patients per month.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven mycosis fungoides/Sezary syndrome Stage I-IV disease No CNS involvement At least 1 measurable lesion required (skin, lymph nodes, visceral lesion, or peripheral blood counts)

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-3 Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 75,000/mm3 Hepatic: Bilirubin no more than 2.0 mg/dL Transaminases no more than 2 x normal Alkaline phosphatase no more than 2 x normal Renal: Creatinine no more than 2.0 mg/dL Other: No active systemic infection No significant organ failure uncontrolled with medication No pregnant or lactating women Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior systemic therapy Chemotherapy: At least 4 weeks since prior topical chemotherapeutics or systemic therapy Endocrine therapy: At least 4 weeks since prior topical (including steroid) therapy or systemic therapy Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1991-10; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Siegel RS, Martone B, Guitart J, et al.: Phase II trial of all-TRA in the treatment of relapsed/refractory mycosis fungoides. 94(1 suppl): A423, 96a, 1999.